CLINICAL TRIAL: NCT05078723
Title: Functional Consequences of CYP2C19 Variants on Limonene Metabolism in Humans
Brief Title: CYP2C19 Variants and Limonene Metabolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Eric Gross, Assistant Professor, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 59978
Record Dates: First submitted 2021-07-01; First posted 2021-10-14 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: CYP2C19 Genetic Variants
MeSH Terms: interventions — Limonene

STUDY DESIGN:
Intervention Model Description: Human volunteers participating in this study will be given an over the counter orange peel extract and limonene levels will be measured.
Masking Description: We are using quantitative assays for this study which reduce the need for masking of the participant or investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CYP2C19*2 and CYP2C19*3 Variants (Experimental): The group of participants has been genotyped to have the CYP2C19*2 and/or CYP2C19*3 variant during the first part of the study. The participants will consume 1 oz water mixed with 500mg limonene (Jarrow Formula orange peel extract) and be asked to swish 5 times and swallow. All participants will then provide breath samples over the course of 2 hours. The breath sample outcomes will be compared to those of the wild-type CYP2C19 study subjects.
  Interventions: Dietary Supplement: Limonene
- Wildtype CYP2C19 (Experimental): The group of participants has been genotyped to have wild-type CYP2C19. The participants will consume 1 oz water mixed with 500mg limonene (Jarrow Formula orange peel extract) and be asked to swish 5 times and swallow. All participants will then provide breath samples over the course of 2 hours. The breath sample outcomes will be compared to those of the CYP2C19*2 and/or CYP2C19*3 study subjects.
  Interventions: Dietary Supplement: Limonene

INTERVENTIONS:
Dietary Supplement: Limonene — The investigators will ask the participants to swish 5 times and swallow 1 oz water mixed with 500mg limonene (Jarrow Formula orange peel extract). The participant will be monitored for a total of 2 hours. Breath samples will be acquired at a total of 11 time points throughout the study. Measurements include 2 baseline measurements followed by the orange peel extract consumption.

SUMMARY:
The investigators will examine whether a non-invasive screening tool for CYP2C19 genetic variants can be developed by measuring limonene metabolism.

DETAILED DESCRIPTION:
Cytochrome P450 2C19 is an important enzyme that metabolizes many drugs. However, individuals with genetic variants of CYP2C19, such as CYP2C19*2 and CYP2C19*3, are poor metabolizers of these drugs. Therefore, it is of interest to determine whether the investigators can develop a non-invasive assay to identify genetic variants of CYP2C19 by using a substrate for CYP2C19 found in citrus fruit, limonene. The purpose of the study is to examine changes in limonene levels in human breath after drinking orange peel extract for people with CYP2C19*2 and CYP2C19*3 genetic variants versus those that do not.

ELIGIBILITY:
Inclusion Criteria:

* Age range: Greater than 18 years and less than 45 years.
* Gender: Male or Female
* Ethnicities: East Asian

Exclusion Criteria:

* Pregnant and/or Breastfeeding
* previous allergic reaction to limonene, citrus fruits, bovine gelatin, glycerin
* past medical history of cerebrovascular or cardiovascular disease
* veganism
* history of chest pain or shortness of breath in the past month
* certain medications that are CYP2C19 substrates or CYP2C19 inhibitors
* Non-East Asian descent
* age less than 18 y.o or age greater than 45 y.o

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Breath limonene value in parts per billion | 2 hours
  The amount of limonene in the breath will be measured by mass spectrometry for each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No